CLINICAL TRIAL: NCT04781569
Title: A Single Centre, Unblinded, Prospective Cohort Study Identifying Pathogen Adaptations in Patients Suffering From Invasive S. Aureus Infection Compared to Colonized, Healthy Individuals
Brief Title: Staphylococcus Aureus Caught in Action at the Site of Infection
Acronym: PROSA
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-00793; me20Khanna
Record Dates: First submitted 2021-02-23; First posted 2021-03-04 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-06

CONDITIONS: Staphylococcus (S.) Aureus Infection
Keywords: antibiotic therapy; virulence factor adaptations; resistance development; genomic alterations of S. aureus
MeSH Terms: interventions — Data Collection; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with S. aureus infection
  Interventions: Other: data collection; Diagnostic Test: blood draw; Diagnostic Test: nose swabs; Diagnostic Test: Intraoperative tissue samples
- healthy participants
  Interventions: Other: data collection; Diagnostic Test: blood draw; Diagnostic Test: nose swabs

INTERVENTIONS:
Other: data collection — Health-related personal data such as year of birth, sex, Body Mass Index (BMI), infection classification, concomitant infections, comorbidities according to medical chart, standard diagnostic markers (CRP, blood differential plots, creatinine, ...), medication, treatment start, treatment end and discharge from hospital will be collected.
Diagnostic Test: blood draw — 2 blood drawing events (in total 22.5 ml) will be performed in the patient. 1 blood drawing events will be performed in the healthy proband.
Diagnostic Test: nose swabs — 2 nose swabs will be taken in the patient. 1 nose swab will be performed in the healthy proband.
Diagnostic Test: Intraoperative tissue samples — Intraoperative tissue samples from the site of infection during surgery will be taken in the patient.
  Groups: Patients with S. aureus infection

SUMMARY:
This study is to obtain a comprehensive view of S. aureus adaptations in the infected human host and (i) to improve the understanding of the interface between antibiotic therapy, resistance development and virulence factor adaptation in S. aureus infected patients, and (ii) to adapt these findings into a more sustainable use of antimicrobials for therapy.

DETAILED DESCRIPTION:
Staphylococcus (S.) aureus is notorious for its ability to develop resistance. This study is to obtain a comprehensive view of S. aureus adaptations in the infected human host and (i) to improve the understanding of the interface between antibiotic therapy, resistance development and virulence factor adaptation in S. aureus infected patients, and (ii) to adapt these findings into a more sustainable use of antimicrobials for therapy.

Patients with S. aureus infections who will routinely undergo diagnostic and surgical procedures will be identified. Intraoperative samples from the site of infection during surgery will be taken. Additionally, two blood drawing events (22.5ml in total) will be performed and nose swabs will be taken. The biological material will be analysed. This project will be the first to study different phenotypes of invasive S. aureus directly from its environment in vivo.

ELIGIBILITY:
Inclusion criteria for patients:

* In collaboration with the orthopedic surgeons, patients with probable or proven S. aureus infections will be identified who will routinely undergo diagnostic and surgical procedures:

Inclusion criteria for healthy participants:

* Healthy control group should be generally well-being

Exclusion criteria for patients and for healthy participants:

* Pregnancy: Pregnant or lactating women will be excluded (urinary pregnancy test will be performed in women of childbearing age)
* General health condition: Current or recurrent disease that could cause complications that may affect the study or may set the patient at risk
* Diseases/ Illness: Psychiatric or other mental disorders which in the opinion of the investigator may probably affect the full understanding of the study (including signs of dementia)
* Language: Insufficient knowledge of german language to understand the procedure and rationale of the research question
* Vulnerability: Individuals whose willingness to volunteer in the research project may be unduly influenced by the expectation, whether justified or not, of benefits associated with participation, such as members of a group with a direct hierarchical structure (refer to ICH Guidelines E6 (R1) for GCP, 1.61)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients with probable or proven S. aureus infection will be screened at the University Hospital of Basel. Patients with confirmed S. aureus infection who correspond to the eligibility criteria will be asked to participate in the research project.
  Healthy volunteers who correspond to the eligibility criteria will be asked to participate in the research project and recruited by oral communication from the institutions Biozentrum, University Hospital Basel, and University of Basel.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-06-06 (Actual); Primary Completion 2020-11-23 (Actual); Study Completion 2020-11-23 (Actual)

PRIMARY OUTCOMES:
Expression of virulence factors of S. aureus (derived from patient's samples (tissue, nose swab)) by combining highly sensitive mass spectrometry with whole genome sequencing. | Project duration for each patient will be two days
  Expression of virulence factors of S. aureus (derived from patient's samples (tissue, nose swab)) by combining highly sensitive mass spectrometry with whole genome sequencing. There is neither a primary nor a secondary endpoint in this research project.
Antibiotics concentration | Project duration for each patient will be two days
  Antibiotics concentration with chromatography methods (in tissue, blood)
Expression of genomic alterations of S. aureus (derived from patient's samples (tissue, nose swab)) by combining highly sensitive mass spectrometry with whole genome sequencing. | Project duration for each patient will be two days
  Expression of genomic alterations of S. aureus (derived from patient's samples (tissue, nose swab)) by combining highly sensitive mass spectrometry with whole genome sequencing. There is neither a primary nor a secondary endpoint in this research project.

CONTACTS AND LOCATIONS:
Overall Officials: Nina Khanna, PD Dr. med., Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland